CLINICAL TRIAL: NCT05359848
Title: A Pilot, Feasibility Study of Intermittent Caloric Restriction Plus Plant-based Protein Diet in Cancer Patients Receiving Chemotherapy
Brief Title: A Pilot, Feasibility Study of Intermittent Caloric Restriction Plus Plant-based Diet in Cancer Patients Receiving Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Roberto Pili, Associate Dean for Cancer Research and Integrative Oncology, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005648
Record Dates: First submitted 2022-04-25; First posted 2022-05-04 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: Medical Oncology; Integrative Oncology; Medical Nutrition Therapy
MeSH Terms: interventions — Diet

STUDY DESIGN:
Intervention Model Description: Patients with cancer where SOC is represented by chemotherapy will be eligible for the study. After informed consent, eligible patients will be scheduled to the chemotherapy. Each cycle will be every 14, 21 or 28 days depending on the regimen. The diet intervention will commence 1 week prior to the first infusion (i.e. on Day -5 for regimens every 21-28 days, on Day-3 for regimens every 14 days) and will continue until the end of cycle 4 or 6 depending on the regimen in the neoadjuvant or adjuvant setting. For metastatic disease the dietary intervention will last until cycle 6 and not beyond
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Diet — Using dietary interventions as an adjuvant tool may represent an effective step toward advancing the treatment options of cancer. Dietary modifications can impact the growth and proliferation of tumors via multiple mechanisms

SUMMARY:
Caloric restriction may alter the response to chemotherapy induced stress response and enhance its antitumor effect. This study intends to use an intermitted caloric restriction protocol with alternate days before the chemotherapy administration to enhance the cytotoxic effect generated by standard treatment of cancer.

DETAILED DESCRIPTION:
This pilot trial will provide preliminary evidence that 1) intermittent caloric restriction and a plant-based diet is feasible in cancer patients; 2) intermittent caloric restriction and a plant-based diet can be safely combined with standard chemotherapy; and 3) intermittent caloric restriction and a plant-based diet may reduce the side effects but increase the antitumor effects of standard chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* • Histologically documented, cancer patients who are eligible to receive cytotoxic chemotherapy.

  * Life expectancy of at least 6 months
  * Adults ≥ 18 years of age
  * Adequate hematologic, renal, and liver function as evidenced by the following:

    * White blood cell (WBC) ≥ 2,500 cells/μL
    * Absolute neutrophil count (ANC) ≥ 1,000 cells/μL
    * Platelet Count ≥ 100,000 cells/μL
    * Hemoglobin (HgB) ≥ 9.0 g/dL
    * Creatinine ≤ 2.0 mg/dL
    * Total bilirubin ≤ 2 x upper limit of normal (ULN)
    * Aspartate aminotransaminase (AST, SGOT) ≤ 2.5 x ULN
    * Alanine aminotransaminase (ALT, SGPT) ≤ 2.5 x ULN

Exclusion Criteria:

* • Eastern Cooperative Oncology Group (ECOG) performance status 2 or higher

  * Treatment with any of the following medications or interventions within 28 days of registration:

    * Systemic corticosteroids; however, use of inhaled, intranasal, and topical steroids is acceptable.
    * High dose calcitriol [1,25(OH)2VitD] (i.e., > 7.0 μg/week)
  * Any infection requiring parenteral antibiotic therapy or causing fever (temperature > 100.5°F or 38.1°C) within 1 week prior to registration
  * A known allergy, intolerance, or medical contraindication to receiving the contrast dye required for the protocol-specified CT/MRI imaging
  * Any medical intervention or other condition which, in the opinion of the Principal Investigator, could compromise adherence with study requirements or otherwise compromise the study's objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
The feasibility of intermittent caloric restriction plus a plant-based diet in cancer patients receiving chemotherapy | 12 Months
  enrollment rate
The feasibility of intermittent caloric restriction plus a plant-based diet in cancer patients receiving chemotherapy | 12 Months
  drop-out rate
The feasibility of intermittent caloric restriction plus a plant-based diet in cancer patients receiving chemotherapy | 12 Months
  compliance with diet measured by self-reports

SECONDARY OUTCOMES:
To obtain preliminary evidence of clinical efficacy of the combination of chemotherapy and intermittent caloric restriction | 12 Months
  objective response rate (partial + complete response)
To obtain preliminary evidence of clinical efficacy of the combination of chemotherapy and intermittent caloric restriction | 12 Months
  progression-free survival (PFS)
To obtain preliminary evidence of clinical efficacy of the combination of chemotherapy and intermittent caloric restriction | 12 Months
  overall survival (OS)

OTHER OUTCOMES:
The safety and tolerability of the combination of chemotherapy and caloric restriction | 12 Months
  assessed using NCI CTCAE

CONTACTS AND LOCATIONS:
Locations (1):
- University at Buffalo / Great Lakes Cancer Care, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided